CLINICAL TRIAL: NCT05522686
Title: The Effect of Different Education Methods Before Invasive Urodynamics on Patients' Anxiety, Pain, Readiness for the Procedure, and Satisfaction Levels: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Different Education Methods Before Invasive Urodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Esra Özden, Principal Investigator and Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Invasive Urodynamics
Record Dates: First submitted 2022-06-11; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Urologic Diseases; Urodynamics
Keywords: pain; anxiety; satisfaction; readiness; patient education; nursing; urodynamics
MeSH Terms: conditions — Urologic Diseases; Pain; Anxiety Disorders; Personal Satisfaction | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients in the Brochure Education Group (Experimental): Patients in the Brochure Education Group were given information about urodynamics in a room reserved for education, and the education brochure was introduced. Patients reviewed the brochure and at the end of the education, it was given to them.
  Interventions: Other: Patients in the Brochure Education Group
- Patients in the Video Education Group (Experimental): Patients in the Video Education Group were informed about urodynamics in a room reserved for education. Patients watched the educational video on a computer. The urodynamics patient education video was shown to patients once during the session. They did not request to watch it again.
  Interventions: Other: Patients in the Video Education Group
- Patients in the Brochure-Supported Video Education Group (Experimental): Patients in the Brochure-Supported Video Education Group were given information about urodynamics in a room reserved for education, and the education brochure was introduced. They examined the brochure and watched the educational video on a computer.
  Interventions: Other: Patients in the Brochure-Supported Video Education Group
- Control Group (Other): Patients in this group were given routine clinical information by the healthcare professional that would perform the urodynamics procedure. After patients were given verbal information, a written text containing the necessary preparations for urodynamics was given to them. The routine patient information text included adjustment to the appointment day and time, nutrition, mechanical bowel preparation, and medications necessary for the procedure.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Patients in the Brochure Education Group — Patients in the Brochure Education Group were given information about urodynamics in a room reserved for education, and the education brochure was introduced. Patients reviewed the brochure and at the end of the education, it was given to them.
  Arms: Patients in the Brochure Education Group
Other: Patients in the Video Education Group — Patients in the Video Education Group were informed about urodynamics in a room reserved for education. Patients watched the educational video on a computer. The urodynamics patient education video was shown to patients once during the session. They did not request to watch it again.
  Arms: Patients in the Video Education Group
Other: Patients in the Brochure-Supported Video Education Group — Patients in the Brochure-Supported Video Education Group were given information about urodynamics in a room reserved for education, and the education brochure was introduced. They examined the brochure and watched the educational video on a computer.
  Arms: Patients in the Brochure-Supported Video Education Group
Other: Control Group — Patients in this group were given routine clinical information by the healthcare professional that would perform the urodynamics procedure. After patients were given verbal information, a written text containing the necessary preparations for urodynamics was given to them. The routine patient information text included adjustment to the appointment day and time, nutrition, mechanical bowel preparation, and medications necessary for the procedure.
  Arms: Control Group

SUMMARY:
Aim: This study was carried out to compare the effects of different education methods utilized before a urodynamic testing procedure on patients' pain, anxiety, readiness for the procedure, and satisfaction.

Background: Urodynamic testing is an invasive procedure that causes pain and anxiety. Patient education is an evidence-based nursing intervention that relieves pain and anxiety and increases patient satisfaction.

Design: The study is a single-center, randomized controlled clinical trial. Method: Participants (n=80) were randomly assigned to four groups. While patients in the control group were provided with routine clinical information, patients in the intervention group were given education with brochures, videos, and brochure-supported videos. The research data were collected by using a Data Collection Form with items about participants' descriptive characteristics, the State Anxiety Inventory, and the Visual Analog Scale.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age,
* Had urodynamics for the first time,
* Had no communication problems,
* Volunteered to participate in the study

Exclusion Criteria:

* Had major hearing, vision, and speech impairments,
* Used antidepressants, or anxiolytic drugs,
* Had an indwelling urinary catheter,
* Used any analgesic in the 24 hours before coming to the urodynamic laboratory

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Anxiety | baseline (before education), pre-urodynamics and immediately after urodynamics
  This is a questionnaire consisting of short statements developed by C.D. Spielberger et al. in 1970. The inventory, which consists of 20 items in total, is used to determine how an individual feels at a certain time and under certain conditions. Scores that can be obtained on the scale range between 20 and 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety (Spielberger, 1983).
Change from Pain | baseline (before education), pre-urodynamics and immediately after urodynamics
  This form, which has three sections, namely pre-education, post-education/pre-procedure, and post-procedure, includes the Visual Analogue Scale (VAS) and a recording table for some physiological parameters (blood pressure, pulse, respiration). The Visual Analogue Scale (VAS) is a valid, reliable, and usable measurement tool for repeated measurements. The VAS has been used in many studies to evaluate readiness for the urodynamic procedure, satisfaction, pain, procedure-related expectation of pain, and willingness to have the procedure again if necessary (Shim, 2017; Warda, 2019; Öztürk, 2019). In this study, readiness for the procedure, satisfaction, procedure-related expectation of pain, and willingness to have the procedure again if necessary, which are among parameters that are thought to affect the subsequent health behaviors of patients, were evaluated by using the VAS.
Change from Readiness for the Procedure | baseline(before education) and pre-urodynamics.
  In this study, readiness for the procedure which are among parameters that are thought to affect the subsequent health behaviors of patients, were evaluated by using the VAS.
Satisfaction management | immediately after urodynamics
  This form, which has three sections, namely pre-education, post-education/pre-procedure, and post-procedure, includes the Visual Analogue Scale (VAS) and a recording table for some physiological parameters (blood pressure, pulse, respiration). The Visual Analogue Scale (VAS) is a valid, reliable, and usable measurement tool for repeated measurements. The VAS has been used in many studies to evaluate readiness for the urodynamic procedure, satisfaction, pain, procedure-related expectation of pain, and willingness to have the procedure again if necessary (Shim, 2017; Warda, 2019; Öztürk, 2019). In this study, readiness for the procedure, satisfaction, procedure-related expectation of pain, and willingness to have the procedure again if necessary, which are among parameters that are thought to affect the subsequent health behaviors of patients, were evaluated by using the VAS.

CONTACTS AND LOCATIONS:
Overall Officials: esra özden, Study Chair — Gulhane Training and Research Hospital
Locations (1):
- Esra Özden, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided